CLINICAL TRIAL: NCT05194345
Title: An Integrated Nutrition Intervention Through the Part C Early Intervention Services to Promote Healthy Eating Habits for Children With ASD
Brief Title: An Integrated Nutrition Intervention to Promote Healthy Eating Habits for Children With ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY002968
Record Dates: First submitted 2022-01-03; First posted 2022-01-18 (Actual); Results first posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Nutrition; Children; Feeding strategies; Intervention
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Data collectors/outcomes assessors will be masked on whether the participants are in the intervention or the control (enhanced usual care) group. 51 parent-child dyads completed the baseline assessments, 50 dyads enrolled (100 individuals) in the intervention/control condition, and 32 providers enrolled to implement the intervention/control. The total number of participants who are considered enrolled is 132 (individuals).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autism Eats nutrition intervention (Experimental): Autism Eats intervention lessons (10 lessons + 2 booster sessions) integrate ASD-specific feeding strategies such as repeated exposures, food chaining, and making regular mealtime routines and behaviorally-focused nutrition content and activities utilizing goal setting, healthy meal planning, monitoring progress, strategies to overcome barriers, and creating healthy home food environment. The early intervention (EI) providers will be trained to implement the lessons. EI providers are well-trained to use personalized intervention and coaching approach in their EI services, which will be applied to Autism Eats activities as well. Each intervention lesson will take 25-30 minutes within one hour EI services, and parent-child dyads will participate in the intervention as part of their regular EI services. The Autism Eats lesson manual will be provided to the EI providers and the parent handbook will be distributed to the parent participants.
  Interventions: Behavioral: Autism Eats nutrition intervention
- We Can! enhanced usual care control (Active Comparator): Enhanced usual care (EUC) control group materials are from the evidence-based materials that are already developed and available online (in both English and Spanish): https://www.nhlbi.nih.gov/health/educational/wecan/index.htm. We will download one to two handouts and email early intervention providers to distribute them to parent-child dyads. Materials will be distributed each week for 10 weeks and additional monthly handouts for two months after the first 10 weeks (parallel to the intervention schedule).
  Interventions: Behavioral: We Can! enhanced usual care

INTERVENTIONS:
Behavioral: Autism Eats nutrition intervention — The Autism Eats intervention group will spend about 8.5 hours over 5 months (baseline, post intervention, and 5-month follow-up assessments are 30 minutes each, 25-30 minutes weekly sessions for up to 10 weeks, two 25-30 minutes monthly booster sessions, and a 60-minute exit interview). The Autism Eats intervention group EI provider will spend about 12 hours over 5 months (two 90-minutes training sessions, 25-30 minutes weekly sessions for up to 10 weeks, two 25-30 minutes monthly booster sessions, 10-minute fidelity checklist completion after each session, and a 60-minute exit interview).
  Arms: Autism Eats nutrition intervention
Behavioral: We Can! enhanced usual care — We Can! EUC control group will spend about 3 hours over 5 months (baseline, post intervention, and 5-month follow-up assessments are 30 minutes each, one 25-30 minute nutrition session, and a 60-minute exit interview). We Can! EUC control group EI provider will spend about 4.5 hours over 5 months (two 90-minutes training sessions, one 25-30 minutes session, 1-2-minute written material distribution at their 9 weekly EI sessions, and a 60-minute exit interview).
  Arms: We Can! enhanced usual care control

SUMMARY:
There is an unmet need for nutrition interventions that address both autism spectrum disorder (ASD) specific feeding challenges and unbalanced eating habits among children with ASD to prevent future chronic health conditions. Children with ASD tend to consume few fruit and vegetables and mainly high-energy dense foods, including sugar-sweetened beverages and processed snacks. Obesity prevalence in children with ASD is up to 40% higher than in typically developing children, and recent studies show significantly elevated risks of hyperlipidemia and hypertension among individuals with ASD, regardless of using psychotropic medications. Our interdisciplinary team conducted a preliminary study to examine diet quality and mealtime behaviors among diverse children with ASD in Florida (34% Hispanic/Latino) and parental preferences for nutrition interventions. Based on the study findings, we developed the manual for our nutrition intervention, Autism Eats, for children with ASD enrolled in the Part C of Individuals with Disabilities Education Act (IDEA) Early Intervention (EI) services. Our Autism Eats manual and parent materials are based on ASD-specific feeding strategies such as food chaining combined with behaviorally-focused nutrition intervention strategies such as goal setting and weekly meal planning to promote healthy eating. Among children with ASD enrolled in Part C EI services in Florida, we will conduct a randomized controlled trial (RCT) with the nutrition intervention program, Autism Eats, and the enhanced usual care (EUC) comparison program. The Autism Eats intervention is to prevent problematic mealtime behaviors and promote development of healthy eating habits. We expect that implementing the Autism Eats will be feasible and the intervention will be well-received by EI providers and parent-child dyads. We will examine differences in children's food intakes (fruit and vegetables), food variety, diet quality, and problematic mealtime behaviors between children in Autism Eats and those in the EUC groups at post-intervention and 5-month follow-up from baseline.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the feasibility and preliminary efficacy of Autism Eats in improving dietary intake and mealtime behaviors of children with ASD. We will enroll 30 early intervention (EI) providers who work with dyads of parent and child with ASD (n=48) and randomly assign them into either the Autism Eats or Enhanced Usual Care (EUC) group. We will test the feasibility of enrollment, implementation, and evaluation of Autism Eats. We expect that Autism Eats will be feasible and well-received by EI providers and parent-child dyads. Feasibility will be determined by benchmarks set in each of the following categories: (1) reach/participation; (2) attrition; (3) completion; (4) fidelity; (5) compatibility; and (6) positive participant feedback. To assess the preliminary efficacy of Autism Eats for improving child dietary intake and mealtime behaviors, we will use a validated tool to assess dietary intake of children and problematic mealtime behaviors. While evaluation of outcomes is more appropriate for a fully-powered clinical trial, we will examine variance and effect sizes of key outcomes at baseline, post-intervention, and 5-month follow-up. We will examine differences in children's food intakes (fruit and vegetables), food variety, diet quality, and problematic mealtime behaviors between children in Autism Eats and those in the EUC groups at post-intervention and 5-month follow-up from baseline. As an exploratory aim, we will explore whether child weight status differs between Autism Eats and EUC groups at 5-month follow-up assessment. Height and weight of children will be measured, and weight-for-length based on the CDC growth chart (birth to 3 years)17 will be calculated and weight status will be determined by the percentile chart by sex. The long-term goal is to identify and implement interventions in early childhood that improve health trajectories in populations with ASD.

Random assignment will be made utilizing a random number generator after baseline data collection is completed. The Autism Eats intervention consists of ten 25-minute weekly lessons, two monthly booster sessions, social media components, and provider training and on-going support. Lessons integrate ASD-specific feeding strategies such as repeated exposures, food chaining, and making regular mealtime routines and behaviorally-focused nutrition content and activities utilizing goal setting, healthy meal planning, monitoring progress, strategies to overcome barriers, and creating healthy home food environment. The EI providers are well-trained to use personalized intervention and coaching approach in their Part C EI services, which will be applied to Autism Eats activities as well (e.g., using the child's favorite foods for lesson activities). Both in-person and telehealth versions of the intervention manual will be available (in case of the COVID-19 pandemic service restriction). There is no content difference between in-person and telehealth versions of the program, except that instructions for providers are tailored to each setting. To maintain scientific control for attention threats and increase rigor, EUC families will also receive a one-time 25-minute session on nutrition and publicly available web-based information on healthy eating (e.g., We Can! materials) weekly over 10-weeks to correspond with the number of Autism Eats sessions. These strategies have been successfully used as comparison offerings in previous RCTs.

The primary outcome measure is dietary intake: food groups, food variety, and diet quality. Data collection times are at baseline, post-intervention (about 10-11 weeks from baseline), and 5-month follow-up from baseline. Three-day food records will be completed by parents and data will be entered into the NCI Automated Self-administered 24-hour Dietary Recall (ASA24) by research assistants. We focus on average daily fruit and vegetables and daily food variety. For all children aged 2 years or older, diet quality will be determined by the Healthy Eating Index's total and sub-component scores (adequacy vs. moderation food categories). There are two secondary outcome measures. The first is problematic mealtime behaviors. The time frame is baseline, post-intervention, and 5-month follow-up from baseline. The Brief Autism Mealtime Behavior Inventory (BAMBI), which is validated and used in many previous research studies will be used to assess children with ASD's problematic mealtime behaviors. Parents will complete the survey via REDCap. The BAMBI contains 18 questions and sues a 5-point scale, with response options ranging from 1 (Never) to 5 (Almost every meal), for reporting the frequency of a behavior. Each question also has a yes or no option for parents to indicate if they perceive the behaviors as problematic. The BAMBI includes the subscales of Limited Variety, Food Refusal, and Features of Autism. The survey takes about 5 minutes to complete. The second is anthropometric- height and weight. The time frame is baseline and 5-month follow-up from baseline. Parents will be given options for their child's and their own anthropometric assessments. They can come to the USF office and get children's and their own height and weight measured by a trained research assistant (RA) or a RA can visit participants' house to use the same portable stadiometer and weight scale. If only virtual height and weight measurement is accessible (due to the COVID-19 pandemic), a metal ruler and a bathroom weight scale will be sent to the participant's house and a RA instructed assessment will be virtually completed. As a standard weight status assessment for birth to 36 months, weight-for-length based on the CDC growth chart will be calculated and weight status will be determined by the percentile chart by sex. Parent BMI will be calculated and used as a covariate in data analyses. If height and weight information is available for the spouse of the participating parent or the other biological father/mother, it will be recorded on the form.

For our RCT, we will enroll a total of 48 parent-child dyads with a randomization between Autism Eats intervention and EUC comparison group. The sample size and power calculation was not formally performed because we do not have our own reference effect size values for the study outcomes and because it is not cost-effective to conduct a full-scale RCT without preliminary data. However, based on our previous studies and literature on calculating preliminary RCT sample sizes, our target sample size of 48 parent-child dyads can be justified. We are using the size of the parent-child dyads because children's dietary behavioral outcomes are the primary RCT outcomes. According to Whitehead et al. (2015) in Statistical Methods in Medical Research journal, pilot RCTs do not have the same objectives as a main trial and using formal power considerations is usually not necessary. We justify our target sample size based on their pilot sample size calculations and recommendations. With an estimated small effect size (0.2), an n=25 pilot RCT sample size (per arm) is recommended. For a medium standardized effect size (0.5), a sample size of 15 per arm is recommended. Based on previous nutrition education literature and from our own experiences, we anticipate seeing a small to medium preliminary effect size (approximately 0.3-0.4) conservatively, and therefore, our sample size of 48 parent-child dyads satisfies their pilot RCT sample size recommendations.

Specific Analyses for the Individual Study Aims: Aim 2a. Test the feasibility of enrollment, implementation, and evaluation of Autism Eats. We hypothesize that Autism Eats will be feasible and well received by EI providers and parent-child dyads, which will be assessed with (1) reach/participation; (2) attrition; (3) completion; (4) fidelity; (5) compatibility; and (6) qualitative feedback from participants. The rates of reach, participation, attrition, and completion will be computed. Descriptive statistics will be used to examine data distributions and frequencies. If there is substantial variability in attrition, completion, fidelity, and compatibility, we will examine the relations of such variables with any other variables we collect during the study such as demographic variables of EI providers and parent-child dyads.

Aim 2b.To assess the preliminary efficacy of Autism Eats on child dietary intake and mealtime behaviors. While evaluation of outcomes is more appropriate for a fully-powered RCT, we will examine variance and effect sizes of key outcomes from pre-to post-intervention, as well as post-intervention to 5-month follow-up using non-parametric tests and confidence intervals. We expect differences in children's food group intakes, variety, diet quality, and mealtime behaviors between children who participate in Autism Eats and those in the EUC groups at post-intervention and 5-month follow-up from baseline. We will first assess whether Autism Eats and EUC groups are balanced through randomization in terms of demographic variables at baseline. For each outcome variable, we will use boxplots and scatterplots with confidence intervals to visually inspect the changes across pre-intervention, post-intervention, and 5-month follow-up by group along with descriptive statistics. Also, nonparametric longitudinal analysis will be conducted for each outcome variable with time as a within-subject factor and treatment condition as a between-subject factor to examine the difference in changes between Autism Eats and EUC groups.

Exploratory Aim. We will explore whether weight status of children are different between Autism Eats and EUC groups at 5-month follow-up assessment. Descriptive statistics and visual inspection will be used to summarize weight status by group and effect sizes will be computed. Similar to the analysis of the primary outcomes, we will conduct nonparametric analysis to compare the changes in weight status at 5-month follow-up between Autism Eats and EUC groups. Note that parent BMI will be included as a covariate in the analysis.

Biological variables. Sex: Given the sex difference in ASD prevalence, in addition to the primary data analyses as described above, data distributions will be analyzed by sex. We will then explore how male and female students respond to our intervention differently through qualitative interviews with selected sub-samples. Recommendations will be created to address any sex differences. Genetic factors: Family history of ASD and parent BMI will be measured and considered as covariates. Potential confounding factors to be considered in the analytic models. Parentage, sex, race/ethnicity, baseline child's weight status, parent education, and family income. Examine demographic variations in response to the Autism Eats intervention. Correlation will be used to examine associations between demographic variations (age, sex, race/ethnicity, SES, and baseline weight status) outcomes of the Autism Eats(food intakes, food variety, diet quality, mealtime behaviors, and weight percentile).

Attrition and Missing Data. We aim <20% dropout due to study withdrawal. Every effort will be made to prevent dropouts/missing data, and to complete relevant assessments for participants who drop out or are withdrawn, including reasons why the intervention was ended. To handle the dropout problem in this trial, we will first analyze data to see whether dropout was related to certain baseline measures and demographic variables. We will report the dropout rate and compare the distributions of baseline measures and demographic variables.

ELIGIBILITY:
Inclusion Criteria:

* Children should be enrolled in the early intervention (EI) service and diagnosed with ASD determined by clinical assessment such as the Autism Diagnostic Observation Schedule (ADOS) or another validated evaluation tool (e.g., Gilliam Autism Rating Scale, GARS-3), if available, or be at-risk/monitored for ASD with a pending diagnosis at the time of screening. Children birth to 36 months are eligible for the EI services, and therefore, age of our research participants will range from birth to 36 months. The ASD diagnosis verification process occurs in two steps: (1) during screening; and (2) at the 5-month follow up assessment, taking into consideration the pending diagnosis at screening and potential changes in diagnosis status due to the young age of the children.
* Both the child and the parent should be available during the EI service time.
* Parents should be 18 years or older and speak fluent English and/or Spanish

Exclusion Criteria:

* Children who are on exclusive breastfeeding, medicines that may interact with appetite and food consumption, having severe GI conditions such as irritable bowel syndrome, diagnosed with feeding disorders or severe food selectivity (consuming fewer than 5 food items), or other serious medical comorbidities such as cancer.
* Children who are receiving the EI service at a daycare setting or other than home setting.
* Parent and child with ASD who have previously participated in a similar nutrition intervention study will also be excluded.
* Parent's first language is not English or Spanish.

Max Age: 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 132 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heewon L Gray, PhD, RDN, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
A study protocol manuscript has been submitted for publication, and all deidentified data will be submitted to the NIH/NIMH NDA system at the end of the study and within a year after the project ends.
Supporting Information: Study Protocol, Analytic Code
Time Frame: A study protocol manuscript has been submitted for publication in Feb 2022, and all deidentified data will be submitted to the NIH/NIMH NDA system at the end of the study and within a year after the project ends.
Access Criteria: Publication on study protocol will be available to public through the journal. Analytic code and deidentified data will be available to those researchers who have permission to use data related to autism spectrum disorder through NIH/NIMH.

REFERENCES:
- [Background] Curtin C, Hyman SL, Boas DD, Hassink S, Broder-Fingert S, Ptomey LT, Gillette MD, Fleming RK, Must A, Bandini LG. Weight Management in Primary Care for Children With Autism: Expert Recommendations. Pediatrics. 2020 Apr;145(Suppl 1):S126-S139. doi: 10.1542/peds.2019-1895P. PMID 32238539
- [Background] Curtin C, Jojic M, Bandini LG. Obesity in children with autism spectrum disorder. Harv Rev Psychiatry. 2014 Mar-Apr;22(2):93-103. doi: 10.1097/HRP.0000000000000031. PMID 24614764
- [Background] Kahathuduwa CN, West BD, Blume J, Dharavath N, Moustaid-Moussa N, Mastergeorge A. The risk of overweight and obesity in children with autism spectrum disorders: A systematic review and meta-analysis. Obes Rev. 2019 Dec;20(12):1667-1679. doi: 10.1111/obr.12933. Epub 2019 Oct 8. PMID 31595678
- [Background] Goldstein BI, Korczak DJ. Links Between Child and Adolescent Psychiatric Disorders and Cardiovascular Risk. Can J Cardiol. 2020 Sep;36(9):1394-1405. doi: 10.1016/j.cjca.2020.06.023. Epub 2020 Jul 3. PMID 32628978
- [Background] Ptomey LT, Walpitage DL, Mohseni M, Dreyer Gillette ML, Davis AM, Forseth B, Dean EE, Waitman LR. Weight status and associated comorbidities in children and adults with Down syndrome, autism spectrum disorder and intellectual and developmental disabilities. J Intellect Disabil Res. 2020 Sep;64(9):725-737. doi: 10.1111/jir.12767. Epub 2020 Jul 27. PMID 32716138
- [Background] Xu G, Strathearn L, Liu B, Bao W. Prevalence of Autism Spectrum Disorder Among US Children and Adolescents, 2014-2016. JAMA. 2018 Jan 2;319(1):81-82. doi: 10.1001/jama.2017.17812. PMID 29297068
- [Background] Xu G, Strathearn L, Liu B, O'Brien M, Kopelman TG, Zhu J, Snetselaar LG, Bao W. Prevalence and Treatment Patterns of Autism Spectrum Disorder in the United States, 2016. JAMA Pediatr. 2019 Feb 1;173(2):153-159. doi: 10.1001/jamapediatrics.2018.4208. PMID 30508021
- [Background] Gray HL, Sinha S, Buro AW, Robinson C, Berkman K, Agazzi H, Shaffer-Hudkins E. Early History, Mealtime Environment, and Parental Views on Mealtime and Eating Behaviors among Children with ASD in Florida. Nutrients. 2018 Dec 2;10(12):1867. doi: 10.3390/nu10121867. PMID 30513809
- [Background] Buro AW, Gray HL, Kirby RS, Berkman K, Agazzi H, Shaffer-Hudkins E. Diet quality in an ethnically diverse sample of children and adolescents with autism spectrum disorder compared with nationally representative data. Disabil Health J. 2021 Jan;14(1):100981. doi: 10.1016/j.dhjo.2020.100981. Epub 2020 Jul 30. PMID 32811783
- [Background] Williams KE, Foxx RM. Treating Eating Problems of children with Autism Spectrum Disorders and Developmental Disabilities Austin, TX: PRO-ED, Inc.; 2007.
- [Background] Contento I. Review of nutrition education research in the Journal of Nutrition Education and Behavior, 1998 to 2007. J Nutr Educ Behav. 2008 Nov-Dec;40(6):331-40. doi: 10.1016/j.jneb.2008.06.001. No abstract available. PMID 18984488
- [Background] Chapman J, Armitage CJ. Evidence that boosters augment the long-term impact of implementation intentions on fruit and vegetable intake. Psychol Health. 2010 Mar;25(3):365-81. doi: 10.1080/08870440802642148. PMID 20204966
- [Background] Fry JP, Neff RA. Periodic prompts and reminders in health promotion and health behavior interventions: systematic review. J Med Internet Res. 2009 May 14;11(2):e16. doi: 10.2196/jmir.1138. PMID 19632970
- [Background] Talbott MR, Dufek S, Zwaigenbaum L, Bryson S, Brian J, Smith IM, Rogers SJ. Brief Report: Preliminary Feasibility of the TEDI: A Novel Parent-Administered Telehealth Assessment for Autism Spectrum Disorder Symptoms in the First Year of Life. J Autism Dev Disord. 2020 Sep;50(9):3432-3439. doi: 10.1007/s10803-019-04314-4. PMID 31776881
- [Background] Stern M, Soca Lozano S, Lescano C, Rodriguez C, Redwine L. Developing Adaptando Dieta Y Accion Para Todos (ADAPT): An Intervention to Improve Healthy Lifestyle Behaviors Among Latino Parents and Children Living in Rural Communities. J Immigr Minor Health. 2021 Feb;23(1):88-94. doi: 10.1007/s10903-020-01037-y. PMID 32533505
- [Background] Lukens CT, Linscheid TR. Development and validation of an inventory to assess mealtime behavior problems in children with autism. J Autism Dev Disord. 2008 Feb;38(2):342-52. doi: 10.1007/s10803-007-0401-5. Epub 2007 Jun 20. PMID 17578658
- [Background] Kuczmarski RJ, Ogden CL, Grummer-Strawn LM, Flegal KM, Guo SS, Wei R, Mei Z, Curtin LR, Roche AF, Johnson CL. CDC growth charts: United States. Adv Data. 2000 Jun 8;(314):1-27. PMID 11183293
- [Background] Maenner MJ, Shaw KA, Baio J; EdS1; Washington A, Patrick M, DiRienzo M, Christensen DL, Wiggins LD, Pettygrove S, Andrews JG, Lopez M, Hudson A, Baroud T, Schwenk Y, White T, Rosenberg CR, Lee LC, Harrington RA, Huston M, Hewitt A; PhD-7; Esler A, Hall-Lande J, Poynter JN, Hallas-Muchow L, Constantino JN, Fitzgerald RT, Zahorodny W, Shenouda J, Daniels JL, Warren Z, Vehorn A, Salinas A, Durkin MS, Dietz PM. Prevalence of Autism Spectrum Disorder Among Children Aged 8 Years - Autism and Developmental Disabilities Monitoring Network, 11 Sites, United States, 2016. MMWR Surveill Summ. 2020 Mar 27;69(4):1-12. doi: 10.15585/mmwr.ss6904a1. PMID 32214087
- [Background] Tyler CV, Schramm SC, Karafa M, Tang AS, Jain AK. Chronic disease risks in young adults with autism spectrum disorder: forewarned is forearmed. Am J Intellect Dev Disabil. 2011 Sep;116(5):371-80. doi: 10.1352/1944-7558-116.5.371. PMID 21905805
- [Background] WHO. Autism spectrum disorders. World Health Organization. https://www.who.int/news-room/fact-sheets/detail/autism-spectrum-disorders. Published 2019. Updated November 7. Accessed October 3, 2020.
- [Background] Burrell TL, Sharp WG, Criado KK, Berry R, Luevano C, Khan R, Scahill L. Feasibility of a Structured, Multidisciplinary Intervention for Weight Management in Children With Autism Spectrum Disorder. Semin Pediatr Neurol. 2020 Oct;35:100830. doi: 10.1016/j.spen.2020.100830. Epub 2020 Jun 23. PMID 32892963
- [Background] Berry RC, Novak P, Withrow N, Schmidt B, Rarback S, Feucht S, Criado KK, Sharp WG. Nutrition Management of Gastrointestinal Symptoms in Children with Autism Spectrum Disorder: Guideline from an Expert Panel. J Acad Nutr Diet. 2015 Dec;115(12):1919-27. doi: 10.1016/j.jand.2015.05.016. Epub 2015 Jul 9. No abstract available. PMID 26164551
- [Background] Evans EW, Must A, Anderson SE, Curtin C, Scampini R, Maslin M, Bandini L. Dietary Patterns and Body Mass Index in Children with Autism and Typically Developing Children. Res Autism Spectr Disord. 2012;6(1):399-405. doi: 10.1016/j.rasd.2011.06.014. PMID 22936951
- [Background] Ledford JR, Gast DL. Feeding Problems in Children With Autism Spectrum Disorders: A Review. Focus on Autism and Other Developmental Disabilities. 2006;21(3):153-166.
- [Background] Mari-Bauset S, Zazpe I, Mari-Sanchis A, Llopis-Gonzalez A, Morales-Suarez-Varela M. Food selectivity in autism spectrum disorders: a systematic review. J Child Neurol. 2014 Nov;29(11):1554-61. doi: 10.1177/0883073813498821. Epub 2013 Oct 4. PMID 24097852
- [Background] Sharp WG, Berry RC, McCracken C, Nuhu NN, Marvel E, Saulnier CA, Klin A, Jones W, Jaquess DL. Feeding problems and nutrient intake in children with autism spectrum disorders: a meta-analysis and comprehensive review of the literature. J Autism Dev Disord. 2013 Sep;43(9):2159-73. doi: 10.1007/s10803-013-1771-5. PMID 23371510
- [Background] Marshall J, Hill RJ, Ziviani J, Dodrill P. Features of feeding difficulty in children with Autism Spectrum Disorder. Int J Speech Lang Pathol. 2014 Apr;16(2):151-8. doi: 10.3109/17549507.2013.808700. Epub 2013 Sep 3. PMID 24001171
- [Background] Curtin C, Hubbard K, Anderson SE, Mick E, Must A, Bandini LG. Food selectivity, mealtime behavior problems, spousal stress, and family food choices in children with and without autism spectrum disorder. J Autism Dev Disord. 2015 Oct;45(10):3308-15. doi: 10.1007/s10803-015-2490-x. PMID 26070276
- [Background] Kral TV, Eriksen WT, Souders MC, Pinto-Martin JA. Eating behaviors, diet quality, and gastrointestinal symptoms in children with autism spectrum disorders: a brief review. J Pediatr Nurs. 2013 Nov-Dec;28(6):548-56. doi: 10.1016/j.pedn.2013.01.008. Epub 2013 Mar 24. PMID 23531467
- [Background] Esteban-Figuerola P, Canals J, Fernandez-Cao JC, Arija Val V. Differences in food consumption and nutritional intake between children with autism spectrum disorders and typically developing children: A meta-analysis. Autism. 2019 Jul;23(5):1079-1095. doi: 10.1177/1362361318794179. Epub 2018 Oct 21. PMID 30345784
- [Background] Bandini LG, Curtin C, Phillips S, Anderson SE, Maslin M, Must A. Changes in Food Selectivity in Children with Autism Spectrum Disorder. J Autism Dev Disord. 2017 Feb;47(2):439-446. doi: 10.1007/s10803-016-2963-6. PMID 27866350
- [Background] Paul C, Williams KE, Riegel K, Gibbons B. Combining repeated taste exposure and escape prevention: an intervention for the treatment of extreme food selectivity. Appetite. 2007 Nov;49(3):708-11. doi: 10.1016/j.appet.2007.07.012. Epub 2007 Aug 7. PMID 17920728
- [Background] Sharp WG, Burrell TL, Jaquess DL. The Autism MEAL Plan: a parent-training curriculum to manage eating aversions and low intake among children with autism. Autism. 2014 Aug;18(6):712-22. doi: 10.1177/1362361313489190. Epub 2013 Oct 7. PMID 24101716
- [Background] Cosbey J, Muldoon D. EAT-UP Family-Centered Feeding Intervention to Promote Food Acceptance and Decrease Challenging Behaviors: A Single-Case Experimental Design Replicated Across Three Families of Children with Autism Spectrum Disorder. J Autism Dev Disord. 2017 Mar;47(3):564-578. doi: 10.1007/s10803-016-2977-0. PMID 27904991
- [Background] Ahearn WH, Castine T, Nault K, Green G. An assessment of food acceptance in children with autism or pervasive developmental disorder-not otherwise specified. J Autism Dev Disord. 2001 Oct;31(5):505-11. doi: 10.1023/a:1012221026124. PMID 11794415
- [Background] Ahearn WH, Kerwin ML, Eicher PS, Shantz J, Swearingin W. An alternating treatments comparison of two intensive interventions for food refusal. J Appl Behav Anal. 1996 Fall;29(3):321-32. doi: 10.1901/jaba.1996.29-321. PMID 8926224
- [Background] Cornish E. Gluten and casein free diets in autism: a study of the effects on food choice and nutrition. J Hum Nutr Diet. 2002 Aug;15(4):261-9. doi: 10.1046/j.1365-277x.2002.00372.x. PMID 12153499
- [Background] Dosman C, Adams D, Wudel B, Vogels L, Turner J, Vohra S. Complementary, holistic, and integrative medicine: autism spectrum disorder and gluten- and casein-free diet. Pediatr Rev. 2013 Oct;34(10):e36-41. doi: 10.1542/pir.34-10-e36. PMID 24085796
- [Background] Elder JH. The gluten-free, casein-free diet in autism: an overview with clinical implications. Nutr Clin Pract. 2008 Dec-2009 Jan;23(6):583-8. doi: 10.1177/0884533608326061. PMID 19033217
- [Background] Herbert MR, Buckley JA. Autism and dietary therapy: case report and review of the literature. J Child Neurol. 2013 Aug;28(8):975-82. doi: 10.1177/0883073813488668. Epub 2013 May 10. PMID 23666039
- [Background] Mulloy A, Lang R, O'Reilly M, Sigafoos J, Lancioni G, Rispoli M. Gluten-free and casein-free diets in the treatment of autism spectrum disorders: A systematic review. Research in autism spectrum disorders. 2010;4(3):328-339.
- [Background] Sathe N, Andrews JC, McPheeters ML, Warren ZE. Nutritional and Dietary Interventions for Autism Spectrum Disorder: A Systematic Review. Pediatrics. 2017 Jun;139(6):e20170346. doi: 10.1542/peds.2017-0346. PMID 28562286
- [Background] Scott-Sheldon LAJ, Hedges LV, Cyr C, Young-Hyman D, Khan LK, Magnus M, King H, Arteaga S, Cawley J, Economos CD, Haire-Joshu D, Hunter CM, Lee BY, Kumanyika SK, Ritchie LD, Robinson TN, Schwartz MB. Childhood Obesity Evidence Base Project: A Systematic Review and Meta-Analysis of a New Taxonomy of Intervention Components to Improve Weight Status in Children 2-5 Years of Age, 2005-2019. Child Obes. 2020 Sep;16(S2):S221-S248. doi: 10.1089/chi.2020.0139. PMID 32936038
- [Background] Hodder RK, O'Brien KM, Tzelepis F, Wyse RJ, Wolfenden L. Interventions for increasing fruit and vegetable consumption in children aged five years and under. Cochrane Database Syst Rev. 2020 May 25;5(5):CD008552. doi: 10.1002/14651858.CD008552.pub7. PMID 32449203
- [Background] Contento IR. Nutrition education: linking research, theory, and practice. Asia Pac J Clin Nutr. 2008;17 Suppl 1:176-9. PMID 18296331
- [Background] Carpenter RA, Finley C, Barlow CE. Pilot test of a behavioral skill building intervention to improve overall diet quality. J Nutr Educ Behav. 2004 Jan-Feb;36(1):20-4. doi: 10.1016/s1499-4046(06)60124-3. PMID 14756978
- [Background] Pivonka E, Seymour J, McKenna J, Baxter SD, Williams S. Development of the behaviorally focused fruits & Veggies--More Matters public health initiative. J Am Diet Assoc. 2011 Oct;111(10):1570-7. doi: 10.1016/j.jada.2011.07.001. PMID 21963025
- [Background] Academy of Nutrition and Dietetics. Pediatric Nutrition Care Manual. https://www.nutritioncaremanual.org/pncm-toc. Accessed March 3, 2019.
- [Background] Gray HL, Contento IR, Koch PA. Linking implementation process to intervention outcomes in a middle school obesity prevention curriculum, 'Choice, Control and Change'. Health Educ Res. 2015 Apr;30(2):248-61. doi: 10.1093/her/cyv005. Epub 2015 Feb 19. PMID 25700557
- [Background] Gray HL, Burgermaster M, Tipton E, Contento IR, Koch PA, Di Noia J. Intraclass Correlation Coefficients for Obesity Indicators and Energy Balance-Related Behaviors Among New York City Public Elementary Schools. Health Educ Behav. 2016 Apr;43(2):172-81. doi: 10.1177/1090198115598987. Epub 2015 Aug 17. PMID 26286297
- [Background] Contento IR, Koch PA, Lee H, Calabrese-Barton A. Adolescents demonstrate improvement in obesity risk behaviors after completion of choice, control & change, a curriculum addressing personal agency and autonomous motivation. J Am Diet Assoc. 2010 Dec;110(12):1830-9. doi: 10.1016/j.jada.2010.09.015. PMID 21111093
- [Background] Contento IR, Koch PA, Lee H, Sauberli W, Calabrese-Barton A. Enhancing personal agency and competence in eating and moving: formative evaluation of a middle school curriculum--Choice, Control, and Change. J Nutr Educ Behav. 2007 Sep-Oct;39(5 Suppl):S179-86. doi: 10.1016/j.jneb.2007.02.006. PMID 17826699
- [Background] Lee H, Contento IR, Koch P. Using a systematic conceptual model for a process evaluation of a middle school obesity risk-reduction nutrition curriculum intervention: choice, control & change. J Nutr Educ Behav. 2013 Mar;45(2):126-36. doi: 10.1016/j.jneb.2012.07.002. Epub 2013 Jan 12. PMID 23321021
- [Background] Majumdar D, Koch PA, Lee H, Contento IR, Islas-Ramos AD, Fu D. "Creature-101": A Serious Game to Promote Energy Balance-Related Behaviors Among Middle School Adolescents. Games Health J. 2013 Oct;2(5):280-290. doi: 10.1089/g4h.2013.0045. PMID 24761326
- [Background] Gray HL, Chiang HM. Brief Report: Mealtime Behaviors of Chinese American Children with Autism Spectrum Disorder. J Autism Dev Disord. 2017 Mar;47(3):892-897. doi: 10.1007/s10803-016-2993-0. PMID 28070790
- [Background] Webber A, Sinha S, Robinson C, Gray HL. Associations Among Diet Variety, Mealtime Behaviors, and Diet Quality in Children with Autism Spectrum Disorder. Journal of Nutrition Education and Behavior. 2018;50(7):S27.
- [Background] Buro A, Gray H. P142 Ethnicity Differences in Nutrient Intake, Diet Quality, and Mealtime Behaviors Among Children with Autism Spectrum Disorder (ASD). Journal of Nutrition Education and Behavior. 2019;51(7):S96
- [Background] Van Arsdale W, Gray H, Buro A. P150 Development of an 8-Week Early Childhood Nutrition Education Intervention for Children with Autism Spectrum Disorder and their Parents. Journal of Nutrition Education and Behavior. 2020;52(7):S87.
- [Background] Families finding the balance: A parent handbook. In: U.S. Department of Health and Human Services NIoH NH, Lung and Blood Institute, ed2005.
- [Background] Mazzeo SE, Kelly NR, Stern M, Gow RW, Cotter EW, Thornton LM, Evans RK, Bulik CM. Parent skills training to enhance weight loss in overweight children: evaluation of NOURISH. Eat Behav. 2014 Apr;15(2):225-9. doi: 10.1016/j.eatbeh.2014.01.010. Epub 2014 Feb 3. PMID 24854808
- [Background] Mazzeo SE, Kelly NR, Stern M, Gow RW, Serdar K, Evans RK, Jones RM, Bulik CM. Nourishing Our Understanding of Role Modeling to Improve Support and Health (NOURISH): design and methods. Contemp Clin Trials. 2012 May;33(3):515-22. doi: 10.1016/j.cct.2012.01.003. Epub 2012 Jan 18. PMID 22273843
- [Background] Stern M, Bleck J, Ewing LJ, Davila E, Lynn C, Hale G, Mazzeo S. NOURISH-T: Targeting caregivers to improve health behaviors in pediatric cancer survivors with obesity. Pediatr Blood Cancer. 2018 May;65(5):e26941. doi: 10.1002/pbc.26941. Epub 2018 Jan 19. PMID 29350459
- [Background] Stern M, Ewing L, Davila E, Thompson AL, Hale G, Mazzeo S. Design and rationale for NOURISH-T: a randomized control trial targeting parents of overweight children off cancer treatment. Contemp Clin Trials. 2015 Mar;41:227-37. doi: 10.1016/j.cct.2014.12.018. Epub 2015 Jan 2. PMID 25559916
- [Background] Steckler A, Linnan L. Process Evaluation for Public Health Interventions and Research. San Francisco, California: Jossey-Bass; 2002.
- [Background] Automated Self-Administered 24-Hour Recall (ASA24). 2011. Published April 25 2017. Accessed October 4, 2014.
- [Background] Zimmer MH, Hart LC, Manning-Courtney P, Murray DS, Bing NM, Summer S. Food variety as a predictor of nutritional status among children with autism. J Autism Dev Disord. 2012 Apr;42(4):549-56. doi: 10.1007/s10803-011-1268-z. PMID 21556968
- [Derived] Gray HL, Jimenez C, Pang T, Kim E, Shaffer-Hudkins E, Agazzi H, Rosado A, Klinger A, Young C, Kandil J, Won S, Perez A, Sayre WD, Waters KA, Miltenberger RG, Stern M. Recruitment feasibility and dietary and behavioral patterns in toddlers with ASD: Preliminary results from the Autism Eats program. Contemp Clin Trials. 2024 Nov;146:107688. doi: 10.1016/j.cct.2024.107688. Epub 2024 Sep 11. PMID 39270747
- [Derived] Gray HL, Pang T, Agazzi H, Shaffer-Hudkins E, Kim E, Miltenberger RG, Waters KA, Jimenez C, Harris M, Stern M. A nutrition education intervention to improve eating behaviors of children with autism spectrum disorder: Study protocol for a pilot randomized controlled trial. Contemp Clin Trials. 2022 Aug;119:106814. doi: 10.1016/j.cct.2022.106814. Epub 2022 Jun 4. PMID 35671902

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One family withdrew due to the participant's own medical reason. Providers were trained and implemented the interventions, but outcomes of the study are assessed mainly for children and some for parents. The target number of providers (n=30 targeted) was met (n=32 enrolled).
Groups:
- Autism Eats Nutrition Intervention: Autism Eats intervention lessons (10 lessons + 2 booster sessions) integrate ASD-specific feeding strategies. The early intervention (EI) providers were trained to implement the lessons. EI providers are well-trained to use personalized intervention and coaching approach in their EI services, which will be applied to Autism Eats activities as well. Each intervention lesson will take 25-30 minutes within one hour EI services, and parent-child dyads will participate in the intervention as part of their regular EI services. The Autism Eats lesson manual will be provided to the EI providers and the parent handbook will be distributed to the parent participants.
  Autism Eats nutrition intervention: The Autism Eats intervention group spent about 8.5 hours over 5 months (baseline, post intervention, and 5-month follow-up assessments are 30 minutes each, 25-30 minutes weekly sessions for up to 10 weeks, two 25-30 minutes monthly booster sessions, and a 60-minute exit interview). The Autism Eats intervention group EI provider spent about 12 hours over 5 months (two 90-minutes training sessions, 25-30 minutes weekly sessions for up to 10 weeks, two 25-30 minutes monthly booster sessions, 10-minute fidelity checklist completion after each session, and a 60-minute exit interview).
- We Can! Enhanced Usual Care Control: Enhanced usual care (EUC) control group materials are from the evidence-based materials that are already developed and available online (in both English and Spanish): https://www.nhlbi.nih.gov/health/educational/wecan/index.htm. Materials were implemented by the EI providers for 10 weeks (weekly, 10 mins per lesson) and additional monthly handouts for two months after the first 10 weeks (parallel to the intervention schedule).
  We Can! enhanced usual care: We Can! EUC control group spent about 3 hours over 5 months (baseline, post intervention, and 5-month follow-up assessments are 30 minutes each, one 25-30 minute nutrition session, and a 60-minute exit interview). We Can! EUC control group EI provider spent about 4.5 hours over 5 months (two 90-minutes training sessions, one 25-30 minutes session, 1-2-minute written material distribution at their 9 weekly EI sessions, and a 60-minute exit interview).
- Providers Trained for Both Intervention and EUC Control: Some providers were trained for both Autism Eats and EUC control programs. The families that they work with were randomly assigned into either group, and the providers were trained for either intervention based on the randomization results.
Period: Overall Study
Arm/Group | Autism Eats Nutrition Intervention | We Can! Enhanced Usual Care Control | Providers Trained for Both Intervention and EUC Control
Started | 64 (25 parent-child dyads (25 parents + 25 children) + 14 providers) | 62 (25 parent-child dyads ((25 parents + 25 children) + 12 providers) | 6 (6 providers who were trained for both Autism Eats and We Can! enhanced usual care control)
Children | 25 | 25 | 0
Parents | 25 | 25 | 0
Providers | 14 | 12 | 6
Completed | 58 (22 parent-child dyads (22 parents + 22 children) + 14 providers) | 56 (22 parent-child dyads (22 parents + 22 children) + 12 providers) | 6
Not Completed | 6 | 6 | 0
Not completed — Withdrawal by Subject | 6 | 4 | 0
Not completed — Moved to another state, becoming ineligible. | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: 25 parent-dyads (50 individuals) per condition: 25 children per condition and 25 parents per condition.
  32 providers implemented the intervention or the enhanced usual care (EUC) control. 14 providers only implemented Autism Eats, 12 providers only implemented EUC, and 6 providers were trained in both programs and implemented the programs based on the random assignments. Outcomes of the providers were not assessed.
Groups:
- Autism Eats Nutrition Intervention: Children: Autism Eats intervention lessons (10 lessons + 2 booster sessions) integrate ASD-specific feeding strategies such as repeated exposures, food chaining, and making regular mealtime routines and behaviorally-focused nutrition content and activities utilizing goal setting, healthy meal planning, monitoring progress, strategies to overcome barriers, and creating healthy home food environment. Each intervention lesson takes 25-30 minutes within one hour EI services, and parent-child dyads participate in the intervention as part of their regular EI services. The Autism Eats intervention group spends about 8.5 hours over 5 months (baseline, post intervention, and 5-month follow-up assessments are 30 minutes each, 25-30 minutes weekly sessions for up to 10 weeks, two 25-30 minutes monthly booster sessions, and a 60-minute exit interview).
- We Can! Enhanced Usual Care Control: Children; We Can! Enhanced Usual Care Control: Parents; We Can! Enhanced Usual Care Control: Providers: Enhanced usual care (EUC) control group materials are from the evidence-based materials that are already developed and available online (in both English and Spanish): https://www.nhlbi.nih.gov/health/educational/wecan/index.htm. Materials were implemented by the EI providers for 10 weeks (weekly, 10 mins per lesson) and additional monthly handouts for two months after the first 10 weeks (parallel to the intervention schedule).
- Autism Eats Nutrition Intervention: Parents: Autism Eats intervention lessons (10 lessons + 2 booster sessions) integrate ASD-specific feeding strategies such as repeated exposures, food chaining, and making regular mealtime routines and behaviorally-focused nutrition content and activities utilizing goal setting, healthy meal planning, monitoring progress, strategies to overcome barriers, and creating healthy home food environment. Each intervention lesson takes 25-30 minutes within one hour EI services, and parent-child dyads participate in the intervention as part of their regular EI services. The Autism Eats lesson manual is provided to the EI providers and the parent handbook is distributed to the parent participants. The Autism Eats intervention group spends about 8.5 hours over 5 months (baseline, post intervention, and 5-month follow-up assessments are 30 minutes each, 25-30 minutes weekly sessions for up to 10 weeks, two 25-30 minutes monthly booster sessions, and a 60-minute exit interview).
- Autism Eats Nutrition Intervention: Providers: Autism Eats intervention lessons (10 lessons + 2 booster sessions) integrate ASD-specific feeding strategies. The early intervention (EI) providers are trained to implement the lessons. EI providers are well-trained to use personalized intervention and coaching approach in their EI services, which are applied to Autism Eats activities as well. Each intervention lesson takes 25-30 minutes within one hour EI services, and parent-child dyads participate in the intervention as part of their regular EI services. The Autism Eats lesson manual is provided to the EI providers and the parent handbook is distributed to the parent participants. The EI providers spend about 12 hours over 5 months (two 90-minutes training sessions, 25-30 minutes weekly sessions for up to 10 weeks, two 25-30 minutes monthly booster sessions, 10-minute fidelity checklist completion after each session, and a 60-minute exit interview).
- Providers Trained for Both Intervention and EUC Control: Some providers were trained for both Autism Eats intervention and EUC control programs and implemented them based on each family's assigned condition.
- Total: Total of all reporting groups
Arm/Group | Autism Eats Nutrition Intervention: Children | We Can! Enhanced Usual Care Control: Children | Autism Eats Nutrition Intervention: Parents | We Can! Enhanced Usual Care Control: Parents | Autism Eats Nutrition Intervention: Providers | We Can! Enhanced Usual Care Control: Providers | Providers Trained for Both Intervention and EUC Control | Total
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 14 | 12 | 6 | 132
Age, Categorical [Count of Participants; unit: Participants]
  Parent (18 and 65 years) and children (<=18 years) dyads: <=18 years | 25 | 25 | 0 | 0 | 0 | 0 | 0 | 50
  Parent (18 and 65 years) and children (<=18 years) dyads: Between 18 and 65 years | 0 | 0 | 25 | 25 | 14 | 12 | 6 | 82
  Parent (18 and 65 years) and children (<=18 years) dyads: >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 25 | 25 | 14 | 12 | 6 | 93
  Male | 19 | 20 | 0 | 0 | 0 | 0 | 0 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 12 | 8 | 12 | 5 | 4 | 4 | 53
  Not Hispanic or Latino | 17 | 13 | 17 | 13 | 9 | 8 | 2 | 79
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
  Asian | 3 | 1 | 3 | 1 | 0 | 0 | 0 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 7 | 3 | 6 | 2 | 1 | 1 | 22
  White | 11 | 12 | 15 | 15 | 7 | 6 | 5 | 71
  More than one race | 9 | 4 | 4 | 2 | 2 | 1 | 0 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 3 | 4 | 0 | 7
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 25 | 25 | 14 | 12 | 6 | 132
Total amount of fruits and vegetables [Mean (Standard Deviation); unit: cup equivalents] — Dietary data were collected through 3-day food records. Data were entered into the ASA24 dietary assessment tool, and food group and nutrient data were generated by the ASA24. Total amount of fruits and vegetables was the daily mean intake of fruits and vegetables in cup equivalents as generated by the ASA24. Population: The mean primary outcome data are only from the children (n=50). Parent data are not collected (n=50). Total amount of fruits and vegetables were collected through 3-day food records. Daily total amount of fruits and vegetables is the mean of those across three days. Therefore, the mean cup equivalents is used as the unit of measure. Cup equivalents is used based on the data generated with the ASA24.
  cup equivalents
    number analyzed (Participants) | 25 | 25 | 0 | 0 | 0 | 0 | 0 | 50
    (all) | 1.5902 (0.9774) | 1.3807 (0.9764) |  |  |  |  |  | 1.4854 (0.9726)

OUTCOME MEASURES:

1. Primary Outcome: Change in Fruit and Vegetable Intake From Baseline, as Measured by the Daily Amount of Fruit and Vegetables Consumed by Children
Description: Change in daily fruit and vegetable intake based on 3-day food records. Daily amount (in cup equivalent) of fruit and vegetable intake from each child participant will be estimated based on parent report 3-day food records. The change amount of fruit and vegetable intake at post- from the baseline and at 5-month follow-up from the baseline will be compared between the intervention and the enhanced usual care (EUC) control groups.
Time Frame: baseline, post-intervention (10 weeks from baseline), and 5-month follow-up
Population: Outcome data were only assessed for children. Mean changes of daily amount of fruits and vegetables were calculated. Daily mean intake was used because the data were collected from 3-day food records. Linear mixed-effects models (LMMs) were conducted using restricted maximum likelihood (REML) estimation to evaluate the effects of the intervention and time interaction on the outcome, adjusting for child age, sex, race, and ethnicity.
Measure: Least Squares Mean (95% Confidence Interval); unit: cup equivalents
Groups:
- Autism Eats Nutrition Intervention: Autism Eats intervention lessons (10 lessons + 2 booster sessions) integrate ASD-specific feeding strategies such as repeated exposures, food chaining, and making regular mealtime routines and behaviorally-focused nutrition content and activities utilizing goal setting, healthy meal planning, monitoring progress, strategies to overcome barriers, and creating healthy home food environment. The early intervention (EI) providers will be trained to implement the lessons. EI providers are well-trained to use personalized intervention and coaching approach in their EI services, which are applied to Autism Eats activities as well. Each intervention lesson takes 25-30 minutes within one hour EI services, and parent-child dyads will participate in the intervention as part of their regular EI services. The Autism Eats lesson manual is provided to the EI providers and the parent handbook is distributed to the parent participants.
  The Autism Eats intervention group spends about 8.5 hours over 5 months (baseline, post intervention, and 5-month follow-up assessments are 30 minutes each, 25-30 minutes weekly sessions for up to 10 weeks, two 25-30 minutes monthly booster sessions, and a 60-minute exit interview). The EI provider spend about 12 hours over 5 months (two 90-minutes training sessions, 25-30 minutes weekly sessions for up to 10 weeks, two 25-30 minutes monthly booster sessions, 10-minute fidelity checklist completion after each session, and a 60-minute exit interview).
Arm/Group | Autism Eats Nutrition Intervention | We Can! Enhanced Usual Care Control
Number analyzed (Participants) | 25 | 25
cup equivalents
  The change amount of fruit and vegetable intake at post- from the baseline | 0.313 [-1.511 to 0.413] | -0.045 [-0.842 to 0.752]
  The change amount of fruit and vegetable intake at 5-month follow-up from the baseline | 0.549 [-0.413 to 1.511] | -0.077 [-1.024 to 0.870]

2. Primary Outcome: Change in Food Variety From Baseline, as Measured by the Daily Food Counts Consumed by Children
Description: Change in daily food counts based on 3-day food records. Daily number of food items from each child participant will be estimated based on parent report 3-day food records. The change in number of daily food items at post- from the baseline and at 5-month follow-up from the baseline will be compared between the intervention and the enhanced usual care (EUC) control groups.
Time Frame: baseline, post-intervention (10 weeks from baseline), and 5-month follow-up
Population: Number of foods from the 3-day food records entered into the ASA24. Food codes in ASA24 represent unique food items, therefore we estimated daily food codes reported on 3-day food records over time. Linear mixed-effects models (LMMs) were conducted using restricted maximum likelihood (REML) estimation to evaluate the effects of the intervention and time interaction on the outcome, adjusting for child age, sex, race, and ethnicity. Least Squared Mean and 95% CI are reported from the output.
Measure: Least Squares Mean (95% Confidence Interval); unit: number of unique food codes per day
Arm/Group | Autism Eats Nutrition Intervention | We Can! Enhanced Usual Care Control
Number analyzed (Participants) | 25 | 25
number of unique food codes per day
  The change in number of foods at post- from the baseline | 0.856 [-1.615 to 3.328] | -0.362 [-2.695 to 1.972]
  The change in number of foods at 5-month follow-up from the baseline | -0.031 [-3.027 to 2.965] | -0.726 [-3.614 to 2.161]

3. Primary Outcome: Change in Diet Quality From Baseline, as Measured by Mean Healthy Eating Index (HEI) Score From the Food Records. HEI Score Ranges From 0 to 100.
Description: Change in HEI score based on 3-day food records. Daily mean HEI score from each child participant will be estimated based on parent report 3-day food records. The change in HEI score at post- from the baseline and at 5-month follow-up from the baseline will be compared between the intervention and the enhanced usual care (EUC) control groups. HEI score ranges 0-100, and higher values represent a better outcome (better diet quality).
Time Frame: baseline, post-intervention (10 weeks from baseline), and 5-month follow-up
Population: Healthy Eating Index (HEI-2015) was calculated based on the 3-day food records. Mean HEI scores were calculated. Linear mixed-effects models (LMMs) were conducted using restricted maximum likelihood (REML) estimation to evaluate the effects of the intervention and time interaction on the outcome, adjusting for child age, sex, race, and ethnicity. Least Squared Mean and 95% CI are reported from the output.
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Autism Eats Nutrition Intervention | We Can! Enhanced Usual Care Control
Number analyzed (Participants) | 25 | 25
scores on a scale
  The change in HEI total score at post- from the baseline | -2.179 [-10.043 to 5.685] | -0.510 [-0.8073 to 7.052]
  The change in HEI total score at 5-month follow-up from the baseline | -1.079 [-10.334 to 8.177] | -0.589 [-9.653 to 8.476]

4. Primary Outcome: Change in Mealtime Behaviors, as Measured by Total Score of the Brief Autism Mealtime Behavior Inventory (Score Ranges 5-90).
Description: The Brief Autism Mealtime Behavior Inventory (BAMBI), which is validated and used in many previous research studies to assess children with ASD's problematic mealtime behaviors. Parents completed the survey via REDCap. The BAMBI contains 18 questions using a 5-point scale, with response options ranging from 1 (Never) to 5 (Almost every meal), for reporting the frequency of a behavior. The total score ranges from 18-90. The higher the score indicated more problematic mealtime behaviors (worse). Each question also has a yes or no option for parents to indicate if they perceive the behaviors as problematic (score range 0-18). There are subscales: Limited Variety, Food Refusal, and Features of Autism. The Limited Variety scale includes 8 items, with a score range of 8-40. The Food Refusal scale has 5 items, with a 5-25 score range. The Features of Autism includes 5 items with a 5-25 score range. The total score is the sum of all scores. The survey takes about 5 minutes to complete.
Time Frame: Baseline, post-intervention (10 weeks from baseline), and 5-month follow-up
Population: The higher score represents more problematic mealtime behaviors. Linear mixed-effects models (LMMs) were conducted using restricted maximum likelihood (REML) estimation to evaluate the effects of the intervention and time interaction on the outcome, adjusting for child age, sex, race, and ethnicity. Least Squared Mean and 95% CI are reported from the output.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Autism Eats Nutrition Intervention | We Can! Enhanced Usual Care Control
Number analyzed (Participants) | 25 | 25
score on a scale
  The change in BAMBI mealtime behavior total scores (range 18-90) at post- from the baseline | -5.151 [-11.353 to 1.051] | -4.268 [-10.691 to 2.154]
  The change in BAMBI mealtime behavior total scores at 5-month follow-up from the baseline | -3.413 [-9.894 to 3.068] | -4.267 [-11.038 to 2.504]
  The change in BAMBI Limited Variety sub-scores (range 8-40) at post- from the baseline | -0.499 [-3.973 to 2.975] | -2.269 [-5.866 to 1.329]
  The change in BAMBI Limited Variety sub-scores (range 8-40) at 5-month follow-up from the baseline | 0.818 [-2.812 to 4.448] | -1.597 [-5.390 to 2.196]
  The change in BAMBI Food Refusal sub-scores (range 5-25) at post- from the baseline | -2.667 [-5.320 to -0.014] | -1.405 [-4.153 to 1.342]
  The change in BAMBI Food Refusal sub-scores (range 5-25) at 5-month follow-up from the baseline | -1.785 [-4.558 to 0.987] | -1.882 [-4.778 to 1.015]
  The change in BAMBI Features of Autism sub-scores (range 5-25) at post- from the baseline | -1.985 [-4.241 to 0.272] | -0.594 [-2.931 to 1.742]
  The change in BAMBI Features of Autism sub-scores (5-25) at 5-month follow-up from the baseline | -2.446 [-4.804 to -0.088] | -0.789 [-3.252 to 1.675]
  The change in BAMBI Number of Problems sub-scores (0-18) at post- from the baseline | -2.831 [-5.893 to 0.232] | -0.056 [-3.227 to 3.115]
  The change in BAMBI Number of Problems sub-scores (0-18) at 5-month follow-up from the baseline | -3.006 [-6.206 to 0.194] | -1.587 [-4.930 to 1.757]

5. Secondary Outcome: Change in Child's Weight-for-length/BMI Percentile (Calculated With Height & Weight), as Measured by Percentile on the CDC Weight-for-length/BMI-for-age Growth Chart.
Description: Parents will be given options for their child's anthropometric assessments. They can come to the USF office and get children's height and weight measured by a trained research assistant (RA) or a RA can visit participants' house to use a portable stadiometer and a weight scale. If only virtual height and weight measurement is accessible (due to the COVID-19 pandemic), a metal ruler and a bathroom weight scale will be sent to the participant's house and a RA instructed assessment will be virtually completed. As a standard weight status assessment for birth to 36 months, weight-for-length percentile for under 2 years and BMI percentile for 2 years or older will be calculated based on the CDC growth chart.
Time Frame: Baseline, 5-month follow-up
Population: Change in WFL or BMI percentile for children with ASD at 5-month follow-up from baseline. Linear mixed-effects models (LMMs) were conducted using restricted maximum likelihood (REML) estimation to evaluate the effects of the intervention and time interaction on the outcome, adjusting for race, and ethnicity. Least Squared Mean and 95% CI are reported from the output.
Measure: Least Squares Mean (95% Confidence Interval); unit: Weight-for-length/BMI percentiles
Arm/Group | Autism Eats Nutrition Intervention | We Can! Enhanced Usual Care Control
Number analyzed (Participants) | 25 | 25
Weight-for-length/BMI percentiles | -10.475 [-29.742 to 8.793] | -2.653 [-23.469 to 18.163]

6. Secondary Outcome: Change in Child Feeding Practices, as Measured in Mean on the Child Feeding Questionnaire Using a 5-point Scale.
Description: Items are measured using a five-point Likert-type scale. Parental beliefs and attitudes regarding child feeding practices are measured in seven domains; perceived responsibility (mean of 3 items), parent perceived weight (mean of 4 items), perceived child weight (mean of 3 items), parents' concerns about child weight (mean of 3 items), monitoring (mean of 3 items), restriction (mean of 8 items), pressure to eat (mean of 4 items). Mean scores of each domain are calculated at each time point. The possible range is 1-5 for all seven domains. High scores represent greater perceived responsibility, higher perceived weight, more concerns about child weight, more feeding practices of monitoring, restriction, and pressure to eat. Higher parental concerns is likely to be associated with more controlling parent feeding practices (higher scores in monitoring, restriction, and pressure to eat), which, in turn, relate to worse/poorer dietary behaviors and health outcomes.
Time Frame: Baseline, 5-month follow-up
Population: Parental feeding practice questionnaire (child feeding questionnaire - CFQ) at 5-month follow-up from baseline. Linear mixed-effects models (LMMs) were conducted using restricted maximum likelihood (REML) estimation to evaluate the effects of the intervention and time interaction on the outcome, adjusting for race, and ethnicity. Least Squared Mean and 95% CI are reported from the output.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Autism Eats Nutrition Intervention | We Can! Enhanced Usual Care Control
Number analyzed (Participants) | 25 | 25
score on a scale
  Change in CFQ Feeding Responsibility subscale scores at post-intervention from baseline | -0.214 [-0.685 to 0.258] | 0.034 [-0.435 to 0.503]
  Change in CFQ Concerns about Child's Weight subscale scores at post-intervention from baseline | -0.299 [-1.131 to 0.532] | -0.484 [-1.310 to 0.343]
  Change in CFQ Restriction subscale scores at post-intervention from baseline | 0.088 [-0.657 to 0.833] | 0.433 [-0.308 to 1.174]
  Change in CFQ Pressure-To-Eat subscale scores at post-intervention from baseline | -0.670 [-1.411 to 0.071] | 0.177 [-0.560 to 0.913]
  Change in CFQ Monitoring subscale scores at post-intervention from baseline | 0.433 [-0.620 to 1.487] | 0.040 [-1.008 to 1.088]
  Change in CFQ Feeding Responsibility subscale scores at 5-month follow-up from the baseline | -0.065 [-0.556 to 0.425] | -0.003 [-0.546 to 0.541]
  Change in CFQ Concerns about Child's Weight subscale scores at 5-month follow-up from the baseline | -.397 [-1.261 to .468] | -.337 [-1.295 to .621]
  Change in CFQ Restriction subscale scores at 5-month follow-up from the baseline | .064 [-.711 to .839] | .140 [-.719 to .998]
  Change in CFQ Pressure-To-Eat subscale scores at 5-month follow-up from the baseline | -.201 [-.971 to .570] | -.087 [-.941 to .766]
  Change in CFQ Monitoring subscale scores at 5-month follow-up from the baseline | .090 [-1.006 to 1.186] | .348 [-.866 to 1.563]

7. Other Pre Specified Outcome: Parent BMI, as Measured in kg/m² Calculated From Height (m) and Weight (kg).
Description: Parent height and weight will be assessed by a trained research assistant or it will be self-reported via REDCap survey. Parent height will be measured with a stadiometer and weight will be measured on a scale. If they are unavailable for assessment, data will be self-reported. Parent BMI (kg/m²) will be calculated and used as a covariate/mediator in data analyses.
Time Frame: Baseline, 5-month follow-up
Population: Change in parent BMI at 5-month follow-up from baseline. Linear mixed-effects models (LMMs) were conducted using restricted maximum likelihood (REML) estimation to evaluate the effects of the intervention and time interaction on the outcome, adjusting for child age, sex, race, and ethnicity. Least Squared Mean and 95% CI are reported from the output.
Measure: Least Squares Mean (95% Confidence Interval); unit: kg/m^2
Arm/Group | Autism Eats Nutrition Intervention | We Can! Enhanced Usual Care Control
Number analyzed (Participants) | 25 | 25
kg/m^2 | .908 [-5.670 to 7.487] | -.987 [-8.259 to 6.285]

ADVERSE EVENTS:
Time Frame: 2 years
Description: Adverse events (e.g., severe malnutrition, accident during the intervention sessions, mental distress, or medical emergency...etc.) were monitored.
Groups:
- We Can! Enhanced Usual Care Control: Children: Enhanced usual care (EUC) control group materials are from the evidence-based materials that are already developed and available online (in both English and Spanish): https://www.nhlbi.nih.gov/health/educational/wecan/index.htm. We will download one to two handouts and email early intervention providers to distribute them to parent-child dyads. Materials will be distributed each week for 10 weeks and additional monthly handouts for two months after the first 10 weeks (parallel to the intervention schedule).
  We Can! enhanced usual care: We Can! EUC control group will spend about 3 hours over 5 months (baseline, post intervention, and 5-month follow-up assessments are 30 minutes each, one 25-30 minute nutrition session, and a 60-minute exit interview). We Can! EUC control group EI provider will spend about 4.5 hours over 5 months (two 90-minutes training sessions, one 25-30 minutes session, 1-2-minute written material distribution at their 9 weekly EI sessions, and a 60-minute exit interview).
Arm/Group | Autism Eats Nutrition Intervention: Children | We Can! Enhanced Usual Care Control: Children | Autism Eats Nutrition Intervention: Parents | We Can! Enhanced Usual Care Control: Parents | Autism Eats Nutrition Intervention: Providers | We Can! Enhanced Usual Care Control: Providers | Providers Trained for Both Intervention and EUC Control
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25 | 0/14 | 0/12 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25 | 0/14 | 0/12 | 0/6
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25 | 0/14 | 0/12 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-10-24): https://cdn.clinicaltrials.gov/large-docs/45/NCT05194345/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-24): https://cdn.clinicaltrials.gov/large-docs/45/NCT05194345/SAP_001.pdf